CLINICAL TRIAL: NCT03813927
Title: Systemic Vitamin D Treatment of Diabetic Patients With Foot Ulcers: a Clinical Controlled Investigation of the Effect on Healing
Brief Title: Vitamin D Treatment of Diabetic Patients With Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: REG-48-2015
Record Dates: First submitted 2019-01-09; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Foot Ulcers; Vitamin D Deficiency
MeSH Terms: conditions — Diabetic Foot; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): supplementation with tablet 170 μg Vitamin D each day.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo, tablet with 20 μg Vitamin D each day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Supplementation with tablet 170 μg Vitamin each day.
  Arms: Vitamin D
Dietary Supplement: Placebo — Placebo with tablet 20 μg Vitamin each day.
  Arms: Placebo

SUMMARY:
The purpose of this study, is to determine whether daily supplements of vitamin D improves wound healing in diabetic patients with chronic foot ulcers.

DETAILED DESCRIPTION:
Project title

"Treatment with oral vitamin D in diabetic patients with chronic foot ulcers on the lower limb; a clinical controlled study of the effect on wound healing".

Abstract

Aims and objectives

The purpose of this study is to determine whether daily supplements of vitamin D improves wound healing in diabetic patients with chronic foot ulcers.

Background

Lifetime risk of developing chronic lower extremity ulcers summarized in type I and type II diabetics is about 25% and the prevalence is approximately 7%. There is often a long term resource consuming disorder where 47% of the diabetic leg and foot ulcers effectively can be treated within 12 months.

In Denmark in 2011 there were more than 300,000 diagnosed type I and type II diabetics, and estimated about 200,000 undiagnosed type II diabetics. Therefore, approximately 35,000 diabetics each year are treated for chronic leg or foot ulcers in the Danish health sector. The treatment of these chronic wounds are associated with significant costs, as well as emotional, physical and financial.

Vitamin D deficiency is a widespread problem, and it is estimated that worldwide there is 1 billion people suffering from vitamin D deficiency. A Danish study from 2012 showed vitamin D deficiency in 52% of adults aged 30 60 years. Vitamin D deficiency is more common in diabetics with chronic foot or leg ulcers, when compared with non diabetics and diabetics without ulcers.

Methods and materials

48 diabetic patients with chronic foot ulcers will be included in the study. The patients will be recruited from the outpatient clinic, department of orthopaedic surgery at Zealand University Hospital, Denmark. The patients will randomly be divided into two groups, respectively treated with vitamin D or placebo.

Expected outcome and perspectives

The investigators expect that this study will show that supplementation with oral vitamin D, will result in a significant effect on wound treatment and healing for a large group of diabetic patients with chronic foot ulcers. This will contribute to a changed procedure in this specific group of patients, leading to measurement of vitamin D status and supplementation with vitamin D if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Diagnosed diabetes.
3. Foot ulcers more than 6 weeks.
4. Informed consent

Exclusion Criteria:

1. Pregnancy
2. Granulomatous diseases such as tuberculosis, sarcoidosis and silicosis
3. Hypercalcemia
4. Supplementation of vitamin D > 20 μg a day
5. Renal disease
6. Liver disease
7. Osteomyelitis
8. Skin cancer.
9. Epilepsy.
10. High blod pressure (> 150/100 mmHg).
11. Indication for surgical revision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Wound healing | 48 weeks or wound healing.
  Wound healing, measured in square cm

SECONDARY OUTCOMES:
Vitamin D blod level status | 48 weeks or wound healing.
  Vitamin D blod level status in intervention Group after supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Max Halschou-Jensen, MD, Study Director — Zeeland University Hospital, Denmark

IPD SHARING:
Plan to Share IPD: Undecided